CLINICAL TRIAL: NCT05916664
Title: Phase II Efficacy Study of a Technology-enabled Care Coaching Service for Families Caring for AD/ADRD
Brief Title: Efficacy Study of Kinto Care Coaching for Dementia Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinto (Industry)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FT001
Record Dates: First submitted 2023-05-11; First posted 2023-06-23 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Alzheimer Disease; Lewy Body Disease; Vascular Dementia; Frontotemporal Dementia; Mixed Dementia
Keywords: Caregiving; Financial Education; Technology; Behavioral Intervention; Caregiver Support Intervention; Financial Literacy; Financial Preparedness; Caregiver Well Being; Caregiver Stress; Caregiver Burden
MeSH Terms: conditions — Dementia; Alzheimer Disease; Lewy Body Disease; Dementia, Vascular; Frontotemporal Dementia; Mixed Dementias; Caregiver Burden

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is a care coaching program that assists caregivers with their general caregiving goals and financial caregiving goals. Caregivers will attend a one-on-one care coaching session conducted via Zoom for 60-75 minutes with a care coach and will engage with their care coach through chat-based interactions after completing the session. If requested, up to two additional care coaching sessions will be scheduled.
  Caregivers also will have the opportunity to attend up to 6 weekly support groups with other caregivers facilitated by a care coach and receive a variety of digital resources through the mobile app.
  Interventions: Behavioral: Kinto Care Coaching
- Control (No Intervention): Control group that does not receive the Caregiver Support Intervention

INTERVENTIONS:
Behavioral: Kinto Care Coaching — Describe the basics of the intervention
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate Kinto's Care Coaching intervention for dementia caregivers.

The main questions it aims to answer are:

Does the intervention help caregivers to address their general caregiving goals Does the intervention help caregivers to address their financial caregiving goals

Participants will have access to:

One-on-one care coaching sessions (via zoom) Up to 6 weekly support groups with other caregivers A variety of digital resources through Kinto's mobile app

Researchers will compare intervention and control groups to see if the program supports caregivers' general and financial caregiving needs.

The efficacy of the intervention also will be examined on key outcomes.

DETAILED DESCRIPTION:
The study will include 300 family caregivers drawn from throughout the US, who will engage remotely with the coaches (and one another) using zoom and Kinto's mobile caregiver app.

Caregivers will be randomly assigned to one of two groups to evaluate the impact of the program by making a comparison of those caregivers who received the program (Group

1) and those caregivers who will not receive the program (Group 2). Caregivers assigned to Group 2, the control condition, will be eligible to receive a modified version of the program after completion of the study and data collection protocols.

The intervention is a care coaching program that assists caregivers with their general caregiving goals and financial caregiving goals. Caregivers will attend a one-on-one care coaching session conducted via Zoom for 60-75 minutes with a care coach and will engage with their care coach through chat-based interactions after completing the session. If requested, up to two additional care coaching sessions will be scheduled.

Caregivers also will have the opportunity to attend up to 6 weekly support groups with other caregivers facilitated by a care coach and receive a variety of digital resources through the mobile app.

As guided by the NIH Stage Model for Behavioral Intervention Development, the primary goal of the Phase 2 study is to examine the efficacy of the program on select outcomes for caregivers (i.e., Stage III Real-World Efficacy). As such, the selected data collection periods of T1 (prior to the intervention), T2 (immediately following the initial six week intervention period) and T3 (45 days following this date) will evaluate the immediate and short-term efficacy of the program.

Recruiting of caregivers is scheduled to begin in May 2023. The study plan targets recruitment of three cohorts, each with one hundred participants. The first intervention group will begin the program in August 2023. Subsequent cohorts will begin the study at 8-9 week intervals. The plan includes a contingency to run two additional cohorts (to mitigate any recruitment or retention risk). In the event that all five cohorts are used to achieve participation goals, the final cohort is scheduled to complete the intervention and survey requirements no later than August of 2024.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

* 18 years or older
* Caring for a family member or close friend with dementia or memory loss
* Providing 5 or more hours of care or support each week
* Not getting paid for the care/support
* Fluent in English, or both Spanish and English
* Living in the United States

They must:

● Have access to a smart phone, reliable internet service and an email address

Exclusion Criteria:

Participants can not:

* Currently be participating in another non-pharmacological intervention
* Have participated in a previous Kinto study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alzheimer's Association Head Office, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between 5/10/23 and 11/30/23. Recruitment and participation in the study occurred remotely.
Groups:
- Intervention: The intervention is a care coaching program that assists caregivers with their general caregiving goals and financial caregiving goals. Caregivers will attend a one-on-one care coaching session conducted via Zoom for 60-75 minutes with a care coach and will engage with their care coach through chat-based interactions after completing the session. If requested, up to two additional care coaching sessions will be scheduled.
  Caregivers also will have the opportunity to attend up to 6 weekly support groups with other caregivers facilitated by a care coach and receive a variety of digital resources through the mobile app.
  Kinto Care Coaching: Describe the basics of the intervention
Period: Overall Study
Arm/Group | Intervention | Control
Started | 249 | 246
Completed | 137 | 192
Not Completed | 112 | 54

BASELINE CHARACTERISTICS:
Population: Baseline participants included those who completed the Time 1 survey and the Time 2 and/or the Time 3 survey/s. For individuals assigned to the intervention condition they needed to have completed the first care coaching session which was set as the minimum required dose for participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 137 | 192 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.57 (12.27) | 53.91 (13.24) | 55.75 (13.04)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 24 | 45 | 69
  Female | 111 | 142 | 253
  Other / Missing | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 28 | 44
  Not Hispanic or Latino | 120 | 161 | 281
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 22 | 37 | 59
  White | 95 | 138 | 233
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 137 | 192 | 329

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Mastery
Description: Caregiver Mastery is a 9-item self-report questionnaire that assesses how competent individuals feel in their role as caregivers of individuals with dementia. Example items include I became more self-confident in providing care and I felt I was pretty good at figuring out what he/she needed. The measure is scored using a 4-point Likert scale (1=strongly disagree to 4=strongly agree) with higher scores indicating greater caregiver mastery. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater caregiver mastery.
Time Frame: Changes in caregiver mastery between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.80 (0.43) | 2.80 (0.47)
  T2 | 3.04 (0.41) | 2.90 (0.45)
  T3 | 3.07 (0.45) | 2.92 (0.43)

2. Primary Outcome: Emotional Health Strain
Description: Emotional Health Strain is a 4-item self-report questionnaire that assesses how emotionally strained individuals feel in their role as caregivers of individuals with dementia. Example items include I was under more stress, strain, or pressure and I was more nervous or bothered by nerves than before. The measure is scored using a 4-point Likert scale (1=strongly disagree to 4=strongly agree) with higher scores indicating more emotional health strain. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater emotional health strain.
Time Frame: Changes in emotional health strain between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.95 (0.78) | 2.86 (0.82)
  T2 | 2.46 (0.85) | 2.64 (0.81)
  T3 | 2.47 (0.87) | 2.67 (0.76)

3. Primary Outcome: Personal Gain
Description: Personal Gain is a 4-item self-report questionnaire that assesses the personal gain experienced by individuals in their role as caregivers of individuals with dementia. Example items include Become more aware of your inner strengths and Become more self-confident. The measure is scored using a 4-point Likert scale (1=not at all to 4=a great deal) with higher scores indicating greater personal gain. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater personal gain.
Time Frame: Changes in personal gain between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.56 (0.84) | 2.53 (0.77)
  T2 | 2.73 (0.84) | 2.54 (0.77)
  T3 | 2.77 (0.82) | 2.55 (0.80)

4. Primary Outcome: Financial Self-Efficacy
Description: Financial Self-Efficacy is a 10-item self-report questionnaire that assesses how efficacious individuals feel in their financial preparedness and skills for managing money as related to their caregiving role. Example items include I am confident that I will be able to successfully manage my loved one's finances and I feel confident in talking with my loved one about their finances. The measure is scored using a 4-point Likert scale (1=not at all to 4=a great deal) with higher scores indicating greater financial self-efficacy. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater financial self-efficacy.
Time Frame: Changes in financial self-efficacy between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.81 (0.60) | 2.77 (0.68)
  T2 | 3.08 (0.63) | 2.87 (0.69)
  T3 | 3.14 (0.64) | 2.97 (0.63)

5. Primary Outcome: ULS-8 Loneliness Scale
Description: The ULS-8 Loneliness Scale is an 11 item self-report questionnaire that assesses how lonely individuals feel with 8 original items and 3 additional items. Example items include I feel very close to one or more people and There are people who really understand me. The measure is scored using a 4-point Likert scale (1=strongly disagree to 4=strongly agree) with lower scores indicating greater feelings of loneliness. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with lower scores indicating greater feelings of loneliness.
Time Frame: Changes in loneliness between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.89 (0.51) | 2.86 (0.52)
  T2 | 2.97 (0.50) | 2.84 (0.52)
  T3 | 2.96 (0.49) | 2.86 (0.58)

6. Primary Outcome: Perceived Financial Knowledge
Description: Perceived Financial Knowledge is a 1-item self-report questionnaire that assesses an individual's perceived knowledge about their financial preparedness and skills for managing money as related to their caregiving role. The item states Please rate your current understanding of how to manage money for you or the person you are caring for. The measure is scored using a 5-point Likert scale (1=no knowledge to 5=expert knowledge) with higher scores indicating greater perceived financial knowledge.
Time Frame: Changes in perceived financial knowledge between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 3.45 (0.93) | 3.42 (0.95)
  T2 | 3.78 (0.83) | 3.55 (0.87)
  T3 | 3.79 (0.84) | 3.59 (0.90)

7. Primary Outcome: Caregiver Burden
Description: Caregiver Burden is a 4-item self-report questionnaire that assesses how much strain and stress individuals feel in their caregiving role for individuals with dementia. Example items include Do you feel that because of the time you spend with your relative that you don't have enough time for yourself and Do you feel stressed between caring for your relative and trying to meet other responsibilities (work/family)? The measure is scored using a 5-point Likert scale (1=never to 5=nearly always) with higher scores indicating greater caregiver burden. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 5, with higher scores indicating greater caregiver burden.
Time Frame: Changes in caregiver burden between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 3.16 (0.79) | 3.23 (0.87)
  T2 | 2.87 (0.85) | 3.05 (0.83)
  T3 | 2.82 (0.86) | 3.10 (0.90)

8. Secondary Outcome: Dyadic Relationship Strain
Description: Dyadic Relationship Strain is a 7-item self-report questionnaire that assesses how strained individuals feel because of their caregiving relationship. Example items include I felt my relationship with him/her was strained and I felt resentful toward him/her. The measure is scored using a 4-point Likert scale (1=strongly disagree to 4=strongly agree) with higher scores indicating greater relationship strain. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater relationship strain.
Time Frame: Changes in relationship strain between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.22 (0.74) | 2.21 (0.70)
  T2 | 1.98 (0.72) | 2.08 (0.66)
  T3 | 2.00 (0.74) | 2.13 (0.71)

9. Secondary Outcome: Role Captivity
Description: Role Captivity is a 3-item self-report questionnaire that assesses the extent to which individuals feel trapped in their role as a caregiver. Example items include I wished I were free to lead my own life and I felt trapped having to care for him/her. The measure is scored using a 4-point Likert scale (1=strongly disagree to 4=strongly agree) with higher scores indicating greater role captivity. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater role captivity.
Time Frame: Changes in role captivity between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.46 (0.86) | 2.41 (0.83)
  T2 | 2.23 (0.84) | 2.38 (0.85)
  T3 | 2.17 (0.84) | 2.38 (0.85)

10. Secondary Outcome: Caregiver Unmet Needs
Description: Caregiver Unmet Needs is a 20-item self-report questionnaire that assesses unmet needs of caregivers. Example items include Do you need more information or help with understanding basic information about dementia? and Ideas to assist with your personal wellbeing as a caregiver? The measure is scored using dichotomous yes/no scoring (1=no/2=yes) with higher scores indicating more unmet needs. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 2, with higher scores indicating more unmet needs.
Time Frame: Changes in unmet needs between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 1.67 (0.21) | 1.70 (0.25)
  T2 | 1.36 (0.26) | 1.56 (0.26)
  T3 | 1.33 (0.27) | 1.52 (0.27)

11. Secondary Outcome: Caregiver Unmet Needs Distress
Description: Caregiver Unmet Needs Distress is a 20-item self-report questionnaire that assesses the resulting distress due to caregiver unmet needs. Example items include How distressing or upsetting is understanding basic information about dementia? and Ideas to assist with your personal wellbeing as a caregiver? The measure is scored using a 4-point Likert scale (1=not distressing to 4=very distressing) with higher scores indicating greater distress due to caregiver unmet needs. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater distress due to caregiver unmet needs.
Time Frame: Changes in unmet needs distress between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.39 (0.59) | 2.45 (0.68)
  T2 | 1.86 (0.57) | 2.29 (0.69)
  T3 | 1.79 (0.58) | 2.18 (0.67)

12. Secondary Outcome: Anxiety
Description: Anxiety is a 7-item self-report questionnaire that assesses symptoms of anxiety. Example items include Feel nervous, anxious or on edge and Feel that you could not stop or control worrying? The measure is scored using a 4-point Likert scale (1=not at all to 4=nearly every day) with higher scores indicating more symptoms of anxiety. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating more symptoms of anxiety.
Time Frame: Changes in anxiety symptoms between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.17 (0.82) | 2.18 (0.81)
  T2 | 1.92 (0.85) | 2.06 (0.79)
  T3 | 1.92 (0.80) | 2.09 (0.78)

13. Secondary Outcome: Depression
Description: Depression is an 11-item self-report questionnaire that assesses symptoms of depression. Example items include Feel depressed and Feel that everything you did was an effort? The measure is scored using a 3-point Likert scale (1=hardly ever to 3=often) with higher scores indicating more symptoms of depression. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 3, with higher scores indicating more symptoms of depression.
Time Frame: Changes in depressive symptoms between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 1.68 (0.44) | 1.73 (0.44)
  T2 | 1.59 (0.43) | 1.71 (0.45)
  T3 | 1.58 (0.43) | 1.70 (0.42)

14. Secondary Outcome: Instrumental and Personal Activities of Daily Living - Difficulty
Description: Instrumental and Personal Activities of Daily Living - Difficulty is a 16-item self-report questionnaire that assesses how much difficulty individuals with dementia experience in completing daily tasks as reported by their caregivers. Example items include How difficult was writing checks, paying bills, or balancing a checkbook? and Preparing a balanced meal? The measure is scored using a 4-point Likert scale (1=not difficult to 4=very difficult) with higher scores indicating more difficulty in completing instrumental activities. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating more difficulty in completing instrumental activities.
Time Frame: Changes in instrumental activities of daily living difficulty between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.48 (0.82) | 2.44 (0.87)
  T2 | 2.49 (0.85) | 2.39 (0.82)
  T3 | 2.55 (0.88) | 2.45 (0.79)

15. Secondary Outcome: Instrumental and Personal Activities of Daily Living - Distress
Description: Instrumental Activities of Daily Living - Distress is a 16-item self-report questionnaire that assesses the resulting distress caregivers experience due to the amount of instrumental activities of daily living difficulty experienced by the individual they care for. Example items include How distressing or upsetting was this for you when the person you care performed these activities: Writing checks, paying bills, or balancing a checkbook? and Preparing a balanced meal? The measure is scored using a 4-point Likert scale (1=not distressing to 4=very distressing) with higher scores indicating greater distress. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater distress.
Time Frame: Changes in instrumental activities of daily living distress between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.08 (0.73) | 2.10 (0.83)
  T2 | 1.95 (0.83) | 2.04 (0.72)
  T3 | 1.93 (0.79) | 2.07 (0.81)

16. Secondary Outcome: Cognition - Difficulty
Description: Cognition - Difficulty is an 8-item self-report questionnaire that assesses how much difficulty individuals with dementia experience with their cognition as reported by their caregivers. Example items include How difficult was remembering recent events? and Knowing what day of the week it is? The measure is scored using a 4-point Likert scale (1=not difficult to 4=very difficult) with higher scores indicating more cognitive difficulty. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating more cognitive difficulty.
Time Frame: Changes in cognitive difficulty between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.65 (0.71) | 2.62 (0.78)
  T2 | 2.52 (0.79) | 2.50 (0.79)
  T3 | 2.60 (0.79) | 2.57 (0.76)

17. Secondary Outcome: Cognition - Distress
Description: Cognition - Distress is an 8-item self-report questionnaire that assesses the resulting distress caregivers experience due to the amount of cognitive difficulty experienced by the person they care for. Example items in reference to the person they are caring for include How distressing or upsetting was this for you: Remembering recent events? and Knowing what day of the week it is? The measure is scored using a 4-point Likert scale (1=not distressing to 4=very distressing) with higher scores indicating greater distress. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater distress.
Time Frame: Changes in cognitive distress between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.02 (0.77) | 2.08 (0.87)
  T2 | 1.82 (0.76) | 1.98 (0.80)
  T3 | 1.85 (0.75) | 2.01 (0.78)

18. Secondary Outcome: Behaviors - Frequency
Description: Behaviors - Frequency is a 14-item self-report questionnaire that assesses the frequency in which individuals with dementia experience dementia-related behaviors as reported by their caregivers. Example items include How often did the person you care for act confused? and Talk or mumble to himself/herself? The measure is scored using a 4-point Likert scale (1=none of the time to 4=most or all of the time ) with higher scores indicating more frequent behaviors. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating more frequent behaviors.
Time Frame: Changes in behavioral frequency between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 2.13 (0.56) | 2.08 (0.60)
  T2 | 1.95 (0.50) | 2.06 (0.55)
  T3 | 2.03 (0.52) | 2.07 (0.50)

19. Secondary Outcome: Behaviors - Distress
Description: Behaviors - Distress is a 14-item self-report questionnaire that assesses the resulting distress caregivers experience due to the behaviors of individuals with dementia. Example items in reference to the person they are caring for include How distressing or upsetting was this for you: Act confused? and Talk or mumble to himself/herself? The measure is scored using a 4-point Likert scale (1=not distressing to 4=very distressing) with higher scores indicating greater distress. The total score (reported in this study) is calculated as the average of the item scores, and ranges from 1 to 4, with higher scores indicating greater distress.
Time Frame: Changes in behavioral distress between the control and intervention conditions will be evaluated across time from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline) and T3 (45 days from T2).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 192
score on a scale
  T1 | 1.98 (0.65) | 1.98 (0.72)
  T2 | 1.73 (0.57) | 1.92 (0.62)
  T3 | 1.84 (0.58) | 1.92 (0.62)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from T1 (baseline) to T2 (post-intervention completion/6-weeks from baseline), and from T2 to T3 (45 days from T2).
Description: The study plan highlighted the potential for (1) caregivers to experience sadness, frustration, or other difficult emotions representing discomfort or risk that is outside of normal daily living for this population, and (2) family caregivers to (i) become extremely distraught or abusive, (ii) unduly monopolize support group time, or (iii) share information that indicates elder abuse and/or financial exploitation. None of these experiences or events occurred during the study.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/192
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/192
Other Adverse Events (participants affected / at risk) | 0/137 | 0/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT05916664/Prot_SAP_000.pdf